CLINICAL TRIAL: NCT07012486
Title: A Pilot Study to Evaluate the Therapeutic Effect of Dihydroartemisinin on Female Androgenetic Alopecia
Brief Title: Efficacy of Dihydroartemisinin for Treating Female Androgenetic Alopecia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2025-112R
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Androgenetic Alopecia (AGA)
Keywords: androgenetic alopecia; dihydroartemisinin
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Active Comparator): oral dihydroartemisinin (DHA) combined with topical minoxidil
  Interventions: Drug: Oral DHA + Topical minoxidil 5%
- Control Arm (Other): topical minoxidil alone
  Interventions: Drug: Topical Minoxidil 5%

INTERVENTIONS:
Drug: Oral DHA + Topical minoxidil 5% — DHA 20mg tid po plus daily topical minoxidil 5% for 180 days
  Arms: Intervention Arm
Drug: Topical Minoxidil 5% — Topical minoxidil 5% daily for 180 days
  Arms: Control Arm

SUMMARY:
The goal of this clinical trial is to learn if dihydroartemisinin (DHA) works to treat Androgenetic Alopecia (AGA) in female adults. The main question it aims to answer is:

• Does DHA increase terminal hair follicles in the vertex area. Researchers will compare oral DHA plus topical minoxidil to topical minoxidil alone in female patients with AGA to see if DHA works to alleviate AGA.

Participants will:

* Receive oral DHA every day plus topical minoxidil or use topical minoxidil alone for 6 months.
* Visit the clinic once every month for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with androgenetic alopecia (AGA)
* No pregnancy plans within the next 6 months

Exclusion Criteria:

* Patients who received systemic medications for hair loss within the past 2 months
* Use of topical medication for hair loss within the past 2 weeks
* Pregnancy or lactation
* Patients with known severe diseases of vital organs (e.g., heart, liver, kidney) or malignancies.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in terminal hair follicles in the vertex area | Baseline and 180-day of treatment
  Terminal hair follicles in the vertex area will be quantified before and at the end of treatment

SECONDARY OUTCOMES:
Change of terminal hair follicle density in the vertex area from baseline to the end of treatment | Baseline and 180-day of treatment
Change of hair density in the vertex area from baseline to the end of treatment | Baseline and 180-day of treatment
Change of terminal hair follicle density in the frontal area from baseline to the end of treatment | Baseline and 180-day of treatment
  Terminal hair follicle density in the frontal area
Change of hair density in the frontal area from baseline to the end of treatment | Baseline and 180-day of treatment
Change of serum total testosterone from baseline to the end of treatment | Baseline and 180-day of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jingjing JIANG, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: After publication
Access Criteria: IPD and supporting information will be avaible to researchers upon reasonable request (e.g. with a practical and meaningful research proposal)